CLINICAL TRIAL: NCT04285944
Title: Operator Radiation Protection During Cardiac Catheterization Using Mavig X-ray Protective Drapes®.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Walter Desmet, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S62469
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Radiation Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Active Comparator)
  Interventions: Other: Mavig X-ray Protective Drapes
- Control (No Intervention)

INTERVENTIONS:
Other: Mavig X-ray Protective Drapes — Mavig X-ray Protective Drapes®
  Arms: Study

SUMMARY:
Interventional cardiologists are exposed to significant doses of scatter radiation during cardiac catheterization and percutaneous coronary intervention. Traditional methods of reducing the radiation dose for operators in the cardiac catheterization laboratory include limiting the use of radiation, radiation protection aprons and shields, and the use of lead eye glasses. Despite these measures several parts of the operators body, including the head and neck, are poorly screened from scatter radiation. Radiation protection drapes have been developed for use in cardiac catheterization but no randomized controlled study has yet been performed with the commercially available Mavig X-ray Protective Drapes®. The aim of this study is to evaluate operator radiation protection using Mavig X-ray Protective Drapes®.

ELIGIBILITY:
Inclusion Criteria:

1. Patient undergoing the procedure is older than 18 years and is planned for a coronary angiogram, cardiac catheterization and/or percutaneous coronary intervention.
2. The coronary angiogram/cardiac catheterization/PCI procedure is elective.
3. The patient undergoing the procedure is male, or if female, has no childbearing potential or is not pregnant.

Exclusion Criteria:

1. The procedure is an emergency and/or the patient is unstable. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Operator radiation dose | Immediate
  Gray

CONTACTS AND LOCATIONS:
Overall Officials: Keir Mccutcheon, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (2):
- Belgium (2):
  - Department of Cardiovascular Disease, University Hospitals Leuven, Leuven
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCutcheon K, Vanhaverbeke M, Dabin J, Pauwels R, Schoonjans W, Desmet W, Bennett J. Efficacy of MAVIG X-Ray Protective Drapes in Reducing CTO Operator Radiation. J Interv Cardiol. 2021 Dec 14;2021:3146104. doi: 10.1155/2021/3146104. eCollection 2021. PMID 34987314
- [Derived] McCutcheon K, Vanhaverbeke M, Pauwels R, Dabin J, Schoonjans W, Bennett J, Adriaenssens T, Dubois C, Sinnaeve P, Desmet W. Efficacy of MAVIG X-Ray Protective Drapes in Reducing Operator Radiation Dose in the Cardiac Catheterization Laboratory: A Randomized Controlled Trial. Circ Cardiovasc Interv. 2020 Nov;13(11):e009627. doi: 10.1161/CIRCINTERVENTIONS.120.009627. Epub 2020 Oct 23. PMID 33092401